CLINICAL TRIAL: NCT00004305
Title: Study of Genetic Anomalies of Complement Related Proteins in Patients With IgA Glomerulonephritis
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Ohio State University (Other)
Other Study IDs: 199/11791; OSU-94H0338
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-04

CONDITIONS: IGA Glomerulonephritis
Keywords: IgA glomerulonephritis; rare disease; renal and genitourinary disorders
MeSH Terms: conditions — Glomerulonephritis, IGA; Rare Diseases; Urogenital Diseases

SUMMARY:
OBJECTIVES: I. Determine whether allelic differences associated with the fourth component of complement, type-1 complement receptor expressed on erythrocytes, and Fc receptor FcgRIII contribute to the pathogenesis of IgA glomerulonephritis (IgA-N).

II. Compare genetic anomalies of these key components in immune complex processing and clearance between juvenile vs adult onset IgA-N vs normal controls.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Participants undergo qualitative genetic analysis of complement-related proteins. Studies include: genomic re-arrangement of 4-gene unit, C4 DNA sequence and RNA expression, type-1 complement receptor DNA sequence, Fc-gamma receptor IIIA isoform analysis, classical and alternative complement activation pathway assays, plasma C4 and C4d protein levels, and immunoglobulin patterns in glomerular deposits.

ELIGIBILITY:
* IgA glomerulonephritis

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105
Dates: Start 1998-01

CONTACTS AND LOCATIONS:
Overall Officials: Lee A. Hebert, Study Chair — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States